CLINICAL TRIAL: NCT00937092
Title: Comparison of High-dose Furosemide Versus the Combination of Low-dose Furosemide and Low-dose Dopamine in Patients With Acute Decompensated Heart Failure
Brief Title: Dopamine in Acute Decompensated Heart Failure (DAD-HF) Trial
Acronym: DAD-HF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Gregory Giamouzis, MD, Department of Cardiology, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUH-DC-101-FT
Record Dates: First submitted 2009-06-29; First posted 2009-07-10 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Acute Heart Failure
Keywords: Heart Failure; Dopamine; Furosemide; Worsening Renal Function; Hypokalemia; Outcomes; Prognosis
MeSH Terms: conditions — Heart Failure; Hypokalemia | interventions — Furosemide; Dopamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-dose furosemide (Active Comparator): High-dose furosemide (HDF): 20 mg/h continuous IV administration for 8 hours
  Interventions: Drug: Furosemide
- low-dose dopamine + low-dose furosemide (Active Comparator): Low-dose furosemide combined with low-dose dopamine (LDFD): continuous IV administration of 5 mg/h furosemide combined with 5 μg/kg/min dopamine for a total of 8 hours
  Interventions: Drug: low-dose dopamine + low-dose furosemide

INTERVENTIONS:
Drug: Furosemide — High-dose furosemide(HDF, furosemide 20 mg/h intravenously)
  Arms: High-dose furosemide
Drug: low-dose dopamine + low-dose furosemide — low-dose furosemide combined with low-dose dopamine (LDFD, furosemide 5 mg/h plus dopamine 5μg/kg/min intravenously)
  Arms: low-dose dopamine + low-dose furosemide

SUMMARY:
The aim of this study is to compare the effects of high-dose furosemide versus low-dose furosemide combined with low-dose dopamine on diuresis, renal function, electrolyte balance, and 60-day post-discharge outcomes in patients hospitalized with acute decompensated heart failure.

DETAILED DESCRIPTION:
Worsening renal function (WRF) and hypokalemia related to diuretic use for acute decompensated heart failure (ADHF) are common and portend poor prognosis. Low dose dopamine infusion improves renal perfusion. Whether dopamine infusion improves diuresis and/or reduces renal complication in ADHF is not known. The aim of this study is to compare the effects of high-dose furosemide (HDF, 40 mg furosemide bolus IV, followed by continuous IV infusion of 20 mg/h for a total of 8 hours) vs. low-dose furosemide combined with low-dose dopamine (LDFD, 40 mg furosemide bolus IV, followed by continuous IV infusion of 5 mg/h furosemide plus 5μg/kg/min dopamine for a total of 8 hours) on diuresis, renal function, electrolyte balance, and 60-day post-discharge outcomes in patients hospitalized with ADHF.

ELIGIBILITY:
Inclusion Criteria:

* patients with New York Heart Association (NYHA) functional class IV heart failure according to the American Heart Association (AHA) classification, namely dyspnea on minimal exertion or rest dyspnea, orthopnea, and paroxysmal nocturnal dyspnea
* signs of congestion (third heart sound or pulmonary rales on physical examination)
* pulmonary congestion on chest x-ray
* serum B-type natriuretic peptide levels > 400 pg/ml or NT-proBNP > 1500 pg/ml
* echocardiographic documentation of systolic or diastolic dysfunction
* all candidate patients must be:
* Age >18 years old
* on medical therapy with an ACE-inhibitor and/or a β-blocker
* experiencing an acute decompensation of known chronic HF
* Having baseline oxygen saturation <90% on admission arterial blood gas

Exclusion Criteria:

* the investigators will exclude patients with:

  * acute de novo HF
  * severe renal failure (serum creatinine > 200 μmol/L or GFR < 30 ml/min/1.73m2)
  * admission systolic blood pressure < 90 mm Hg
  * severe valvular disease
  * known adverse reactions to furosemide or dopamine
  * HF secondary to congenital heart disease
  * a scheduled procedure with a need for IV contrast dye
  * a scheduled cardiac surgery within 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
1-year mortality or rehospitalization (all-cause, cardiovascular, non-cardiovascular, and due to worsening heart failure). | 1-year

SECONDARY OUTCOMES:
60-day mortality or rehospitalization (all-cause, cardiovascular, non-cardiovascular, and due to worsening heart failure). | 60 days post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Giamouzis, MD, Principal Investigator — Larissa University Hospital; Filippos Triposkiadis, MD, Principal Investigator — Larissa University Hospital
Locations (2):
- Greece (2):
  - Department of Cardiology, Larissa University Hospital, Larissa, Larissa
  - Department of Cardiology, Volos General Hospital, Volos, Magnesia

REFERENCES:
- [Derived] Giamouzis G, Butler J, Starling RC, Karayannis G, Nastas J, Parisis C, Rovithis D, Economou D, Savvatis K, Kirlidis T, Tsaknakis T, Skoularigis J, Westermann D, Tschope C, Triposkiadis F. Impact of dopamine infusion on renal function in hospitalized heart failure patients: results of the Dopamine in Acute Decompensated Heart Failure (DAD-HF) Trial. J Card Fail. 2010 Dec;16(12):922-30. doi: 10.1016/j.cardfail.2010.07.246. PMID 21111980